CLINICAL TRIAL: NCT00508040
Title: Evaluation of Birdshot RETINE CHOROIDOPATHY Treatment by Either Steroid or Interferon alpha2a
Acronym: BIRDFERON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P051032
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2008-10

CONDITIONS: Birdshot Chorioretinopathy; Cystoid Macular Edema; Transient Partial Visual Loss
Keywords: Birdshot Retine choroidopathy; Macular edema; Prednisone; Interferon alpha 2a; Associated with Cystoid macular edema; With Visual acuity loss
MeSH Terms: conditions — Birdshot Chorioretinopathy; Macular Edema | interventions — Interferon alpha-2; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): To analyse the potential therapeutic effect of Interferon alpha2a versus Steroid therapy with a control group for a 4 months period. This short period could not expose to a worsening of the disease because of the slow pathologic processus.
  Interventions: Drug: interferon alpha 2a; Drug: prednisone
- B (Active Comparator)
  Interventions: Drug: interferon alpha 2a; Drug: prednisone

INTERVENTIONS:
Drug: interferon alpha 2a — We propose to analyse the potential therapeutic effect of Interferon alpha2 a versus Steroid therapy with a control group for a 4 months period. This short period could not expose to a worsening of the disease because of the slow pathologic processus.
Drug: prednisone — We propose to analyse the potential therapeutic effect of Interferon alpha2 a versus Steroid therapy with a control group for a 4 months period. This short period could not expose to a worsening of the disease because of the slow pathologic processus.

SUMMARY:
Birdshot Retine choroidopathy (BRC) is a sight threatening posterior uveitis. The long term visual outcome has recently be studied showing a legal blindness to 14% at 5 years. Visual acuity is threatened by macular edema (80%), macular atrophy, and choroidal neovascularization.

DETAILED DESCRIPTION:
Birdshot Retine choroidopathy (BRC) is a sight threatening posterior uveitis. The long term visual outcome has recently be studied showing a legal blindness to 14% at 5 years. Visual acuity is threatened by macular edema (80%), macular atrophy, and choroidal neovascularization.

The conventional therapy includes in first line steroid therapy of which side effects are well known. If the daily steroid dose necessary to control the intra ocular inflammation is superior to 0.3 mg/kg/d a combined therapy to immunosuppressive drug is suggested in order to do a steroid sparing effect. Immunosuppressive drugs include increased infectious risks, hematologic and sterility troubles, and secondary malignancies. Moreover immunosuppressive drugs have a own toxic effect and The classical immunosuppressive drug used in BRC the cyclosporineA has a high level of nephrotoxicity.

That is the reason why immunomodulatory drugs as interferons have been suggested in BRC.

Interferon alpha2 a has been shown efficient in uveitis in Behcet's disease. We propose to analyse the potential therapeutic effect of Interferon alpha2 a versus Steroid therapy with a control group for a 4 months period. This short period could not make the disease worse because of the slow pathologic processus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Birdshot Retine choroidopathy with macular edema
* HLA A29 positive
* Work up of infection or sarcoidosis disease negative

Exclusion Criteria:

* Pregnancy
* Alcohol addiction
* Mood disturbance
* Medullar, hepatic, renal deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-09; Primary Completion 2011-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Decreasing in macular-center thickness measured with optical coherence tomography | during 4 months

SECONDARY OUTCOMES:
Increasing in best corrected visual acuity | at 4 months and at the end of the study
Final best corrected visual acuity in ETDRS scale | at the 4 month and at the end of the study
Retinal vessels inflammation in fluorescein angiography | at the 4 month and at the end of the study
Choroidal inflammation in indocyanine green angiography | at the 4 month and at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Christine FARDEAU, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital La Pitie Salpetriere, Paris, France

REFERENCES:
- [Result] Kotter I, Gunaydin I, Zierhut M, Stubiger N. The use of interferon alpha in Behcet disease: review of the literature. Semin Arthritis Rheum. 2004 Apr;33(5):320-35. doi: 10.1016/j.semarthrit.2003.09.010. PMID 15079763